CLINICAL TRIAL: NCT05606952
Title: Color Doppler to Confirm Epidural Catheter Positioning in Parturient, Would it Help
Brief Title: Color Doppler to Confirm Epidural Catheter Positioning in Parturient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/2022ANET1-2
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (C) (Active Comparator): patients with BMI less than 35
  Interventions: Device: Color Doppler
- Group (O) (Active Comparator): patients with BMI more than 35
  Interventions: Device: Color Doppler

INTERVENTIONS:
Device: Color Doppler — color Doppler with pulsed wave Doppler to accurately detect the position of epidural catheter
  Other Names: Epidural catheter

SUMMARY:
The aim of this study is to calculate the sensitivity and specificity of using color Doppler with pulsed wave Doppler to accurately detect the position of epidural catheter

DETAILED DESCRIPTION:
patients will be divided into two groups Group (C) control these are the patients with BMI less than 35 and Group (O) for patients with BMI more than 35.All patients will be sitting to receive their epidural analgesia for labor pain.

A 2.5 to 5 MHz curvilinear probe (Sonosite X-porte, Fujifilm industries) will be used to detect the desired level usually between L3-4 or L4-5. patients will be divided into two groups Group (C) control these are the patients with BMI less than 35 and Group (O) for patients with BMI more than 35. All patients will be sitting to receive their epidural analgesia for labor pain.

A 2.5 to 5 MHz curvilinear probe (Sonosite X-porte, Fujifilm industries) will be used to detect the desired level usually between L3-4 or L4-5. Initially a parasagittal oblique interlaminar view will be obtained and by tilting it medially to visualize the laminae and interlaminar spaces. Starting by the sacral image, counting will start detecting the L5-S1, L4-L5 and L3-L4 levels. After marking the level another imaging in the transverse view will be attempted at the previous levels then the anesthetist will detect the posterior complex (ligamentum flavum, epidural space and dura) and anterior epidural complexes and according to the anesthetist preference a level will be This is followed by a test dose of 10 ml 0.125% bupivacaine and patient controlled epidural analgesia will be started by the following protocol (0.0625% bupivacaine) Smith Medical ASD,Inc. in intermittent dose (10 ml will be injected by the machine every 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* obstetric patients admitted for epidural analgesia in the labor department suite (LDS)

Exclusion Criteria:

1. Patients suffering from coagulopathy.
2. Patients on recent anticoagulant therapy.
3. Patients suffering from sepsis or with local sepsis at the insertion site.
4. Patients with platelet count less than 100,000/dl.
5. Patient refusal.
6. Patient with known allergy to local anesthetic drugs
7. Patients delivered by forceps.
8. Patients who have undergone a cesarean section delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Labour analgesia
Enrollment: 194 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
sensitivity | 30 min
  Number and percentage of patients in both groups where the flow was detected

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Menoufia, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No